CLINICAL TRIAL: NCT02454244
Title: Efficacy of Amygdala Retraining With Mindfulness (ART+MF) vs Compassion Therapy (CT) for the Treatment of Patients With Fibromyalgia: A Three-arm Randomized, Controlled Trial.
Brief Title: Efficacy of Amygdala Retraining With Mindfulness (ART+MF) vs Compassion Therapy (CT) for the Treatment of Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Medicine, Psychiatry, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI15/0049
Record Dates: First submitted 2015-05-18; First posted 2015-05-27 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amygdala Retraining Technique (ART) with Mindfulness (Experimental): Consists of 10 weekly sessions, followed by 3 monthly sessions
  Interventions: Behavioral: ART with Mindfulness
- Mindfulness Compassion (Experimental): Includes the attentional training aspect of mindfulness and meditation practices, proved to bring benefits in relation to fibromyalgia and CFS symptoms, as fatigue and pain. Compassion training focuses on the ability to be kind to participants and their own experience, specifically to their experience of suffering. The protocol consists of 10 weekly sessions, followed by 3 following monthly sessions
  Interventions: Behavioral: Mindfulness Compassion
- Relaxation (Active Comparator): Consists of 10 weekly sessions, followed by 3 monthly sessions
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: ART with Mindfulness — 1. Introduction of ART with Mindfulness. Visualization of 100% recovery
  2. Developing Fibromyalgia and CFS. How stress triggers the central nervous system. The benefits of Mindfulness in chronic stress. Mindfulness Practice. Breathing meditation
  3. The ART. Breaking the negative thoughts related to the illness. Walking meditation
  4. Mindfulness and the Body Scan. Breaking the cycle of stress. Body-scan meditation
  5. Mindfulness and self-compassion. Kindly awareness meditation
  6. The accelerator of ART. Behaviors related to CFS and Fibromyalgia. Metta meditation
  7. Aware of negative thoughts related to stress stimulus. Mindfulness in daily activities
  8. Limiting beliefs, identity patterns. Motivation and sense of life. Meditation on values
  9. The recovery, cycles and stages. Fear of fail about recovery. Positive Visualization of future self
  10. Return to regular life. Mindfulness practice
  Arms: Amygdala Retraining Technique (ART) with Mindfulness
Behavioral: Mindfulness Compassion — 1. Introduction.Definition of Compassion
  2. Self-Esteemed and Compassion
  3. Cultivate the understanding of the nature of inner experience. Working positive and negative thoughts.Connecting with difficult emotions
  4. Identifying the causes of suffering.How participants contribute to their own suffering. Attachments.Practice of Vulnerability
  5. Love,affection and self-compassion.How participants connect with the suffering of others
  6. Equanimity
  7. Forgiveness
  8. Interdependence. Gratitude.Affection to unknown people
  9. Developing affection and empathy.Empathy and burn out
  10. Review of the practices and meditations
  Arms: Mindfulness Compassion
Behavioral: Relaxation — 10 sessions based on relaxation techniques as active comparator intervention
  Arms: Relaxation

SUMMARY:
Amygdala Retraining Treatment (ART) is a new and promising therapy for patients with Chronic Fatigue Syndrome (CFS) and Fibromyalgia (FM), however, randomized controlled trials (RCT) are scarce. The investigators have added mindfulness to this therapy, based on preliminary reports of its efficacy on patients, obtaining Amygdala Retraining Treatment with Mindfulness (ART+MF).

Other therapy that has been assessed in many psychiatric and medical disorders during the last years has been Compassion Therapy (CT). There are no studies on its efficacy in FM.

Aims: The aim of this trial is to assess the efficacy of both ART+MF and CT on the general function of the patients with FM. A secondary objective is to assess the effect of these therapies on psychological (pain, depression, anxiety, etc.) and biological variables (some biomarkers related with inflammation).

Methods:

* Design: Randomized, controlled trial with three arms: a) ART+MF, b) CT and c) Relaxation as control intervention.
* Sample: A sample (N=60 patients, about N=20 for each arm) will be recruited from primary care settings at the city of Zaragoza, Spain.

ELIGIBILITY:
Inclusion criteria

1. Male or female aged between 18-65 years.
2. The patient needs to have the ability to read and understand Spanish
3. All the patients included in the study have been diagnosed with FM by a rheumatologist working for the Spanish National Health Service.
4. It is required that the patient does not modify during the trial the pharmacological treatment prescribed.
5. Signed informed consent.

Exclusion criteria

The patient should not meet any of the following criteria during the study:

1. Age <18 years or> 65 years.
2. The patients considered for exclusion are individuals with severe axis I psychiatric disorders (dementia, schizophrenia, paranoid disorder, alcohol and/or drug use disorders) and with severe somatic disorders that, from the clinician's point of view, prevented patients from carrying out a psychological assessment or participating in other clinical trials
3. It is not considered an exclusion criterion antidepressant use, as long as the treatment is not modified during the study period (treatment can be decreased, never increased).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | baseline
Change post-intervention (3 months) Fibromyalgia Impact Questionnaire (FIQ) | post-intervention (3 months)
Change follow-up (6 months) Fibromyalgia Impact Questionnaire (FIQ) | follow-up (6 months)

SECONDARY OUTCOMES:
Sociodemographic Data | baseline
Hospital Anxiety and Depression Scale (HADS) | baseline
Change post-intervention (3 months) Hospital Anxiety and Depression Scale (HADS) | post-intervention (3 months)
Change follow-up (6 months) Hospital Anxiety and Depression Scale (HADS) | follow-up (6 months)
Fibrofatigue Scale (FFS) | baseline
Change post-intervention (3 months) Fibrofatigue Scale (FFS) | post-intervention (3 months)
Change follow-up (6 months) Fibrofatigue Scale (FFS) | follow-up (6 months)
Euroqol Quality of Life Questionnaire | baseline
Change post-intervention (3 months) Euroqol Quality of Life Questionnaire | post-intervention (3 months)
Change follow-up (6 months) Euroqol Quality of Life Questionnaire | follow-up (6 months)
Pain Catastrophizing Scale | baseline
Change post-intervention (3 months) Pain Catastrophizing Scale | post-intervention (3 months)
Change follow-up (6 months) Pain Catastrophizing Scale | follow-up (6 months)
Acceptance Questionaire AAQ-II | baseline
Change post-intervention (3 months) Acceptance Questionaire AAQ-II | post-intervention (3 months)
Change follow-up (6 months) Acceptance Questionaire AAQ-II | follow-up (6 months)
Five Facets Mindfulness Questionaire FFMQ | baseline
Change post-intervention (3 months) Five Facets Mindfulness Questionaire FFMQ | post-intervention (3 months)
Change follow-up (6 months) Five Facets Mindfulness Questionaire FFMQ | follow-up (6 months)
Self-compassion Scale | baseline
Change post-intervention (3 months) Self-compassion Scale | post-intervention (3 months)
Change follow-up (6 months) Self-compassion Scale | follow-up (6 months)
Serum Levels of Interleukins IL-6, IL-10 | baseline
Change post-intervention (3 months) Serum Levels of Interleukins IL-6, IL-10 | post-intervention (3 months)
Serum levels of Brain Derived Neurotrophic Factor BDNF | baseline
Change post-intervention (3 months) Serum levels of Brain Derived Neurotrophic Factor BDNF | post-intervention (3 months)
High-sensitivity C-reactive Protein | baseline
Change post-intervention (3 months) High-sensitivity C-reactive Protein | post-intervention (3 months)
Serum levels of Tumor Necrosis Factor TNF alpha | baseline
Change post-intervention (3 months) Serum levels of Tumor Necrosis Factor TNF alpha | post-intervention (3 months)

REFERENCES:
- [Derived] Montero-Marin J, Andres-Rodriguez L, Tops M, Luciano JV, Navarro-Gil M, Feliu-Soler A, Lopez-Del-Hoyo Y, Garcia-Campayo J. Effects of attachment-based compassion therapy (ABCT) on brain-derived neurotrophic factor and low-grade inflammation among fibromyalgia patients: A randomized controlled trial. Sci Rep. 2019 Oct 30;9(1):15639. doi: 10.1038/s41598-019-52260-z. PMID 31666651
- [Derived] Montero-Marin J, Navarro-Gil M, Puebla-Guedea M, Luciano JV, Van Gordon W, Shonin E, Garcia-Campayo J. Efficacy of "Attachment-Based Compassion Therapy" in the Treatment of Fibromyalgia: A Randomized Controlled Trial. Front Psychiatry. 2018 Jan 16;8:307. doi: 10.3389/fpsyt.2017.00307. eCollection 2017. PMID 29387020